CLINICAL TRIAL: NCT00573859
Title: The Reinforcing Mechanisms of Smoking in Adult ADHD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 2006-5156; NIH grant# DA018752
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Results first posted 2011-11-07 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2011-09

CONDITIONS: ADHD
Keywords: Smoking; ADHD; Stimulant medication
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Smoking | interventions — Dextroamphetamine; Atomoxetine Hydrochloride; Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ADHD medication versus placebo (Experimental): For the ADHD medication condition, participants received their usual dosage of their usual ADHD medication (e.g., Dextroamphetamine; Amphetamine mixed salts; Atomoxetine; O-Methylphenidate; Lisdexamfetamine). For the placebo condition, a placebo pill was administered.
  Interventions: Drug: ADHD medication; Drug: Placebo

INTERVENTIONS:
Drug: ADHD medication — For the ADHD medication condition, participants received their usual dosage of their usual ADHD medication for two consecutive days.
  Other Names: Dextroamphetamine; Amphetamine mixed salts; Atomoxetine; O-Methylphenidate; Lisdexamfetamine
Drug: Placebo — For the placebo condition, participants received placebo pills for two consecutive days.

SUMMARY:
Whereas the smoking prevalence rates in the general population are declining, rates among people diagnosed with attention-deficit hyperactivity disorder (ADHD) continue to be elevated. Smoking may be a form of self-medication in people with ADHD, which has specific reinforcing mechanisms such as improvement of ADHD core symptoms, enhancement of moods and arousal, or a combination of both. In addition, the reinforcing effects of smoking may be potentiated by stimulant medication.

The study examined the reinforcing effects of ad libitum smoking with and without ADHD medication in adult smokers with clinically diagnosed ADHD. Participants were adults with ADHD. The effects of two day of ADHD medication compared to two days on placebo for were studied on nicotine intake (i.e., cotinine levels). In addition, task performance on the Continuous Performance Task and nicotine withdrawal symptoms were examined in response to ADHD medication + smoking a cigarette versus ADHD medication + abstinence versus placebo medication + smoking versus placebo medication + abstinence.

The study identified the reinforcing mechanisms of smoking in interaction with ADHD medication. The findings will contribute to a better understanding of nicotine addiction and facilitate the development of targeted smoking cessation and prevention programs for individuals with ADHD and other people with deficiencies in impulse control and excessive risk taking.

ELIGIBILITY:
Inclusion Criteria:

* An age of 18 to 45 years
* A history of ADHD
* Current diagnosis of ADHD according to clinical criteria
* Current treatment with stimulant medication
* Smoking of 10 cigarettes or more per day

Exclusion Criteria:

* Treatment for any major medical illness such as cancer, heart disease, diabetes, skin diseases, current major depressive episode, and schizophrenia even if currently controlled by medication
* Current pregnancy, as measured by a pregnancy test (Clear Blue Easy, Unipath, Bedford, UK), or planning to become pregnant within the next 6 months. These individuals will not be included because smoking may cause harm to the unborn fetus
* Nursing mothers
* Non-English speaking people, because the majority of measurements used in the study have not been validated in languages other than English

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2006-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean G Gehricke, Ph.D., Principal Investigator — University of California, Irvine
Locations (1):
- Department of Pediatrics, Irvine, California, United States

REFERENCES:
- [Result] Gehricke JG, Hong N, Wigal TL, Chan V, Doan A. ADHD medication reduces cotinine levels and withdrawal in smokers with ADHD. Pharmacol Biochem Behav. 2011 May;98(3):485-91. doi: 10.1016/j.pbb.2011.02.021. Epub 2011 Feb 26. PMID 21356232

RESULTS

PARTICIPANT FLOW:
Groups:
- ADHD Medication Versus Placebo: Smokers with ADHD participated in two consecutive days under ADHD medication versus 2 consecutive days on placebo. For the ADHD medication condition, participants received their usual dosage of their usual medication in the morning of each monitoring day. For the placebo condition, a placebo pill was provided in the morning of each day. The smoking period assessed the effects of the first cigarette of the day on secondary outcome measures. The abstinence period assessed the effects of overnight abstinence on the secondary outcome measures.
Period: Medication Versus Placebo
Arm/Group | ADHD Medication Versus Placebo
Started | 27
Completed | 15
Not Completed | 12
Not completed — Scheduling conflicts | 12
Period: Smoking Versus Abstinence
Arm/Group | ADHD Medication Versus Placebo
Started | 27
Completed | 15
Not Completed | 12
Not completed — Scheduling conflicts | 12

BASELINE CHARACTERISTICS:
Arm/Group | ADHD Medication Versus Placebo
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 27.2 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: The Effects of ADHD Medication Versus Placebo on Cotinine Levels
Description: Salivary cotinine was measured across two days on ADHD medication versus two days on placebo.
Time Frame: 4 days
Population: Smokers with ADHD
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | ADHD Medication Versus Placebo
Number analyzed (Participants) | 15
ng/ml
  ADHD medication | 180.7 (33.3)
  Placebo | 274.0 (70.4)
Statistical Analysis 1: Comparison: ADHD Medication Versus Placebo; A 2 (ADHD medication versus Placebo) repeated measure ANOVA; Test type: Superiority or Other; p < 0.05, ANOVA

2. Secondary Outcome: The Interacting Effects of Smoking and Overnight Abstinence With ADHD Medication and Placebo on Continuous Performance Task (CPT) Errors of Omission.
Description: In the morning of each monitoring day, approximately 60 minutes after medication or placebo pill administration, participants were asked to either abstain from smoking or smoke their first cigarette of the day 5 minutes prior to starting the CPT.
Time Frame: 4 days
Measure: Mean (Standard Error); unit: errors
Arm/Group | ADHD Medication Versus Placebo
Number analyzed (Participants) | 15
errors
  ADHD medication + Smoking | 0.40 (0.1)
  ADHD medication + Abstinence | 1.08 (0.3)
  Placebo + Smoking | 1.00 (0.4)
  Placebo + Abstinence | 2.8 (0.6)
Statistical Analysis 1: Comparison: ADHD Medication Versus Placebo; Four-way repeated measure ANOVA; Test type: Superiority or Other; p < 0.05, ANOVA

3. Secondary Outcome: The Interacting Effects of Smoking and Abstinence With ADHD Medication and Placebo on Nicotine Withdrawal Measured by the Shiffman-Jarvik Withdrawal Questionnaire.
Description: The Shiffman-Jarvik withdrawal questionnaire measures nicotine withdrawal and was completed after each CPT assessment. The questionnaire consists of 25 items using 8-point scales. Total scores range from 0 to 200 and higher scores reflect higher levels of nicotine withdrawal.
Time Frame: 4 days
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | ADHD Medication Versus Placebo
Number analyzed (Participants) | 15
scores on a scale
  ADHD medication + Smoking | 92.7 (2.9) [75 to 123]
  ADHD medication + Abstinence | 91.3 (3.5) [68 to 132]
  Placebo + Smoking | 97.0 (4.8) [59 to 137]
  Placebo + Abstinence | 102.0 (4.8) [80 to 161]
Statistical Analysis 1: Comparison: ADHD Medication Versus Placebo; Friedman's two-way analysis of variance by ranks; Test type: Superiority or Other; p < 0.05, Friedman's two analysis of ranks

ADVERSE EVENTS:
Arm/Group | ADHD Medication Versus Placebo
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No